CLINICAL TRIAL: NCT04095390
Title: A Phase Ⅱ Trial Program Exploring The Integration Of Novel HER2-targeted Tyrosine Kinase Inhibitor Pyrotinib and CDK4/6 Inhibitor SHR6390 Into Current Chemotherapy/Endocrine Therapy Regimes For Prior Trastuzumab-treated Advanced HER2-positive Breast Cancer
Brief Title: A Phase Ⅱ Trial of Pyrotinib Combination With CDK4/6 Inhibitor SHR6390 in Patients Prior Trastuzumab-treated Advanced HER2-Positive Breast Cancer
Acronym: INPHASE
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Jinming Yu (Other)
Collaborators: Jiangsu HengRui Medicine Co., Ltd. (Industry)
Responsible Party: Sponsor-Investigator, Jinming Yu, Director of Shandong Cancer Hospital and Institute, Shandong Cancer Hospital and Institute
Organization: Shandong Cancer Hospital and Institute (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HR-BLTN-010
Record Dates: First submitted 2019-09-16; First posted 2019-09-19 (Actual); Last update posted 2019-09-19 (Actual); Status verified 2019-09

CONDITIONS: Metastatic Breast Cancer; HER2-positive Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — pyrotinib; Letrozole; Capecitabine

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Arm A (Experimental): Hormone receptor positive,HER2 positive participants will receive Pyrotinib in combination with CDK4/6 Inhibitor SHR6390 plus Letrozole until disease progression, unacceptable toxicity, withdrawal of consent or death, whichever occurs first.
  Interventions: Drug: Pyrotinib; Drug: SHR6390; Drug: Letrozole
- Arm B (Experimental): Hormone receptor negative,HER2 positive participants will receive Pyrotinib in combination with CDK4/6 Inhibitor SHR6390 plus Capecitabine until disease progression, unacceptable toxicity, withdrawal of consent or death, whichever occurs first.
  Interventions: Drug: Pyrotinib; Drug: SHR6390; Drug: Capecitabine
- Arm C (Experimental): Hormone receptor negative,HER2 positive participants will receive Pyrotinib in combination with CDK4/6 Inhibitor SHR6390 until disease progression, unacceptable toxicity, withdrawal of consent or death, whichever occurs first.
  Interventions: Drug: Pyrotinib; Drug: SHR6390

INTERVENTIONS:
Drug: Pyrotinib — 400 mg
Drug: SHR6390 — 125mg
Drug: Letrozole — 2.5mg
  Arms: Arm A
Drug: Capecitabine — 500mg
  Arms: Arm B

SUMMARY:
The study is being conducted to evaluate the efficacy, safety and tolerability of pyrotinib combination with CDK4/6 Inhibitor SHR6390 in advanced HER2-Positive breast cancer patients who prior trastuzumab-treated.

ELIGIBILITY:
Inclusion Criteria:

1. Metastatic HER2-Positive breast cancer prior trastuzumab-treated;
2. 18-70 Years, female;
3. HER2-positive breast cancer(according to 2018 ASCO/CAP HER2 test guideline IHC 3+ or IHC 2+ and FISH, SISH or CISH+);
4. Status of hormone receptor is known, Estrogen receptor(ER) or Progesterone receptor(PR) positive is defined as the percentage of cells positive for ER or PR expression ≥ 10%;
5. ECOG performance status 0 or 1;
6. Life expectancy is not less than 12 weeks;
7. At least one measurable lesion according to RECIST 1.1;
8. Patients treated with systemic treatment for advanced / metastatic breast cancer≤1 line;
9. Natural postmenopausal or OFS in Arm A;
10. Adequate function of major organs meets the following requirements (no blood components have been used within 7 days and cell growth factors have been used within 14 days before randomization):

    * Neutrophils ≥ 1.5×10^9/L
    * Platelets ≥ 100×10^9/L
    * Hemoglobin ≥ 90g/L
    * Total bilirubin≤ 1.5 × the upper limit of normal (ULN)
    * ALT and AST ≤ 2.5 × ULN (ALT and AST≤5×ULN if liver metastasis)
    * BUN and Cr ≤ 1.5 × ULN
    * Left ventricular ejection fraction (LVEF) ≥ 50%
    * QTcF ≤ 470 ms

Exclusion Criteria:

1. Patients with central nervous system metastasis (Excluding asymptomatic brain metastases or CNS metastases stable by local treatment);
2. Unable to swallow, chronic diarrhea and intestinal obstruction, gastrointestinal absorption disorders that interfere with drug absorption;
3. Patients who received radiotherapy, chemotherapy, surgery (excluding local puncture) or molecular targeted therapy within 4 weeks before admission; those who received anti-tumor endocrine therapy after screening period;
4. Participated in other drug clinical trials within 4 weeks before admission;
5. Tyrosine kinase inhibitors targeting HER2 (Neratinib, Lapatinib, pyrotinib, etc.) have been used or are being used in the past;
6. Previously received any CDK4/6 inhibitor treatment;
7. Previously received Capecitabine in HR- patients;
8. Patients with other malignant tumors within 5 years or at the same time( except for cured skin basal cell carcinoma and cervical carcinoma in situ);
9. Patients receive any anti-tumor treatments other than the regimen;
10. Have a history of allergies to the drug components of this regimen,; history of immunodeficiency, including HIV positive, or other acquired or congenital immunodeficiency disease, history of organ transplantation;
11. Have severe heart disease;
12. According to the judgement of the researchers, any serious coexisting disease might be harmful to the patient's safety or avoid the patients from accomplishing the treatment(e.g serious hypertension, diabetes, thyroid dysfunction,active infection etc.);
13. Female patients during pregnancy and lactation, fertile women with positive baseline pregnancy tests or women of childbearing age who are unwilling to take effective contraceptive measures throughout the trial;
14. History of neurological or psychiatric disorders, including epilepsy or dementia;
15. Any other situation evaluated by researchers.

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2019-09-30 (Estimated); Primary Completion 2021-11-30 (Estimated); Study Completion 2022-08-30 (Estimated)

PRIMARY OUTCOMES:
Objective Overall Response Rate (ORR) | 2 months
  ORR was defined as percentage of participants with best (confirmed) overall response (BOR) of either CR or PR. ORR was assessed by the investigator according to RECIST version 1.1 and is based on BOR, which is defined as best response recorded from start of study treatment until disease progression/recurrence or death. Participants needed to have two consecutive assessments of PR or CR to be a responder. Only participants with measurable disease at baseline were included in the analysis of BOR and who did not have any evaluable post-baseline assessments were classified as not evaluable.
  The ORR will be reported by percentage with each arms and appropriate confidence intervals.

SECONDARY OUTCOMES:
Progression-Free Survival (PFS) | Up to 3 years
  PFS was defined as the time from randomization to first documented disease progression (PD) using Response Evaluation Criteria in Solid Tumors 1.1 (RECIST 1.1) or death from any cause, whichever occurred first.
Overall Survival (OS) | Up to 3 years
  Overall Survival (OS), defined as the time from the date of randomization to the date of death, regardless of the cause of death. Participants who were alive at the time of the analysis were censored at the date of the last follow-up assessment. Participants without follow-up assessment were censored at the day of last study medication and participants with no post-baseline information were censored at the date of randomization.
Survival Rate | 12 months
  Survival rate was defined as the time from randomization to 12month, the rate of participants who were alive at the time in total.
Clinical Benefit Response (CBR) | 2 months
  CBR is percentage of participants with best (confirmed) PR or CR or SD for at least 6 months. PR or CR or SD is according to RECIST version 1.1.
Adverse Events (AEs) | Up to 3 years
  AEs were graded according to the National Cancer Institute's Common Toxicity Criteria for Adverse Events (CTCAE) version 5.0.
  In general, AEs are graded according to the following: Grade 1 Mild AE Grade 2 Moderate AE Grade 3 Severe AE Grade 4 Life-threatening or disabling AE Grade 5 Death related to AE.
  The type, grade and frequency of AEs will be reported.

CONTACTS AND LOCATIONS:
Locations (1):
- Breast Cancer Center, Shandong Cancer Hospital Affiliated to Shandong University, Jinan, China